CLINICAL TRIAL: NCT06595160
Title: Determining the Link Between Dietary Patterns, Fecal Microbiome and Response to Neoadjuvant Chemotherapy in Pancreatic Ductal Adenocarcinoma Patients
Brief Title: Determining the Link Between Dietary Patterns, Fecal Microbiome and Response to Neoadjuvant Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mihir M. Shah, MD, FACS, FSSO, Principal Investigator, Emory University
Other Study IDs: STUDY00007728; NCI-2024-06743 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00007728 (Other Grant/Funding Number: Emory University Hospital/Winship Cancer Institute); EU6255-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Borderline Resectable Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Ductal Adenocarcinoma; Stage I Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Shotgun Sequencing - Fecal Specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete a dietary survey and undergo fecal sample collection on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study explores the relationship between pre-treatment dietary patterns, fecal microbiome, and response to chemotherapy in patients with pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the association between pre-treatment diversity of the fecal microbiome and major pathological response to neoadjuvant chemotherapy in operable pancreatic ductal adenocarcinoma patients.

II. Evaluate the association between pre-treatment HEI-2015 dietary score and major pathological response to neoadjuvant chemotherapy in pancreatic ductal adenocarcinoma patients.

III. Evaluate the association between pre-treatment HEI-2015 dietary score and diversity of the fecal microbiome in pancreatic ductal adenocarcinoma patients.

OUTLINE: This is an observational study.

Patients complete a dietary survey and undergo fecal sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* * Age ≥ 18 years with signed informed consent form

  * Patients must have a histological diagnosis of PDAC
  * Resectable or borderline resectable PDAC on imaging

Exclusion Criteria:

* * Patients with locally advanced and metastatic stage IV PDAC

  * Patients who have already received or completed neoadjuvant chemotherapy for PDAC
  * Patients with active malignancy receiving systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resectable or borderline resectable pancreatic ductal adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
Fecal Microbiome Alpha Diversity | Through study completion, an average of two years
  Continuous variables will be presented as median with interquartile range and categorical variables will be presented as frequencies. Univariate logistic regression will be used to compare alpha diversity (mean inverse Simpson index) and relative abundance of operational taxonomic units up to species level in PDAC patients with and without major pathological response to neoadjuvant chemotherapy. Multivariable logistic regression analyses will be performed to identify significant factors associated with major pathological response after adjusting for age, gender, stage at presentation, and type of neoadjuvant chemotherapy and other factors based on univariate analyses or clinical significance.

SECONDARY OUTCOMES:
Pathological Response Rate | Through study completion, an average of two years
  Major pathological response rate in surgical specimen of operable PDAC patients after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mihir M Shah, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States